CLINICAL TRIAL: NCT05555693
Title: Correlation Between Postoperative Cognitive-related Adverse Reactions and Brain Metabolomic Characteristics in Elderly Patients
Status: Recruiting | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Other Study IDs: SH9H-2022-T133-2
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: POCD - Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients in the control group were followed up without POCD postoperatively.: If the MOCA or MMSE assessment all show a negative resluts at all time point.
  Interventions: Other: Collecting clinical data, EGG，Brain Metabolomic Characteristics(with Magnetic Resonance Spectroscopy), blood gas data and blood sample
- Patients in the case group were followed up with POCD postoperatively.: If the MOCA assessment is positive at any time point after surgery, and there is a positive MMSE at any time point after surgery(no need for both MOCA and MMSE to be positive at the same time
  Interventions: Other: Collecting clinical data, EGG，Brain Metabolomic Characteristics(with Magnetic Resonance Spectroscopy), blood gas data and blood sample

INTERVENTIONS:
Other: Collecting clinical data, EGG，Brain Metabolomic Characteristics(with Magnetic Resonance Spectroscopy), blood gas data and blood sample — Collecting clinical data(before induction of anesthesia and first day after surgery), EGG（first day after surgery），Magnetic Resonance Spectroscopy data (before induction of anesthesia and first day after surgery)blood gas data(before induction of anesthesia and first day after surgery) and blood sample （before induction of anesthesia and first day, third day and 7th day after surgery）

SUMMARY:
Postoperative cognitive dysfunction (POCD) refers to the difficulties of orientation, cognition, communication, memory and abstract thinking of patients after anesthesia and surgery. And/or accompanied by the decline of the ability in social activities, such as the change of personality, social ability of language and behavior, cognitive function and life skills. POCD is a common complication of central nervous system in elderly patients after operation, with an early incidence of about 21% and a long-term incidence of about 35% . According to the current research on Alzheimer's disease (AD) and POCD in the elderly, it has been found that they have similar pathological basis and some homologous related genes. Altogether, POCD is closely related to molecular pathway neuropsychiatric diseases (such as dementia, depression and Alzheimer's disease). Researchers have come up with various hypotheses to reveal the underlying mechanisms of POCD, including neuritis, oxidative stress, autophagy disorder, synaptic dysfunction, and lack of neurotrophic support. To date, apart from evaluating with scales, CT Scan and EEG analysis, there is neither exact biomarkers for monitoring and diagnosing POCD, nor clear relationships between specific Brain Metabolomic Characteristics, EEG changes and diagnosis of POCD, so that the diagnosis of early POCD only stays in the evaluation of clinical symptoms and scales. Therefore, our study aims to provide an effective basis for early diagnosis and treatment of clinical POCD through multivariate analyses of clinical scales combined with Brain Metabolomic Characteristics, EEG analysis of patients.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older .
* Complete the operation in our hospital
* ASA classification I-II level
* Agree to participate in this research and agree to sign an informed consent form

Exclusion Criteria:

* History of preoperative psychosis and psychotropic drug use
* The subject is diagnosed with AD;
* Abnormal preoperative mental scale assessment
* Have a history of emergency rescue during the perioperative period
* metal implants
* Postoperative immobilization patients

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Our research is a single center, nested case-control study. Preoperatively collect the information of the elderly patients over 65 years old without undergoing craniocerebral operations, including the vital signs, the examination reports and other related data after excluding the factors that can't be included in the group. The patients' health scales and preoperative cognitive function scales were evaluated.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
MMSE (mini-mental state examiniation) | 1 day after surgery
  MMSE scale score, If the MMSE assessment is positive at any time point, and there is a positive MMSE at any time point (no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of POCD.
MMSE (mini-mental state examiniation) | immediately before surgery
  MMSE scale score, If the MMSE assessment is positive at any time point, and there is a positive MMSE at any time point (no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of POCD.
MMSE (mini-mental state examiniation) | 3 day after surgery
  MMSE scale score, If the MMSE assessment is positive at any time point, and there is a positive MMSE at any time point (no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of POCD.
MMSE (mini-mental state examiniation) | 7 day after surgery
  MMSE scale score, If the MMSE assessment is positive at any time point, and there is a positive MMSE at any time point (no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of POCD.
MOCA (Montreal Cognitive Assessment) | 1 day after surgery
  MOCA sacle score, If the MOCA assessment is positive at any time point, and there is a positive MMSE at any time point (no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of POCD.
MOCA (Montreal Cognitive Assessment) | 3 day after surgery
  MOCA sacle score, If the MOCA assessment is positive at any time point, and there is a positive MMSE at any time point (no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of POCD.
MOCA (Montreal Cognitive Assessment) | 7 day after surgery
  MOCA sacle score, If the MOCA assessment is positive at any time point, and there is a positive MMSE at any time point (no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of POCD.
MOCA (Montreal Cognitive Assessment) | immediately before surgery
  MOCA sacle score, If the MOCA assessment is positive at any time point, and there is a positive MMSE at any time point (no need for both MOCA and MMSE to be positive at the same time), it is defined as the occurrence of POCD.

SECONDARY OUTCOMES:
3D-CAM | 1 day after surgery
  3D-CAM score
Self-Rating Anxiety Scale | immediately before surgery
  Self-Rating Anxiety Scale score
Self-rating depression scale | immediately before surgery
  Self-rating depression scale score

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai 9Th Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No